CLINICAL TRIAL: NCT01654198
Title: FDG-PET/CT in the Diagnosis and Monitoring of Psoriatic Arthritis
Brief Title: PET/CT in Psoriatic Arthritis
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 815253
Record Dates: First submitted 2012-07-27; First posted 2012-07-31 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, Serum, and Plasma Cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Psoriatic arthritis
  Interventions: Radiation: FDG-PET/CT scan

INTERVENTIONS:
Radiation: FDG-PET/CT scan — FDG-PET/CT is a type of imaging used currently to look for cancer. We are using it to look at inflammation within the joints.

SUMMARY:
When patients with psoriasis develop joint pain, it is often hard to decide whether or not the pain is due to psoriatic arthritis (PsA). At this time, doctors use information from the history and physical exam to determine the diagnosis. X-rays, magnetic resonance imaging (MRI) and ultrasound have been used to help with the diagnosis but all three have limitations. A newer imaging technique, whole body Positron Emission Tomography/Computed Tomography (PET/CT) uses the idea that inflammatory cells take up sugar to locate inflammation in the body. Because patients with PsA have inflammatory cells in their joints and tendons, this type of scan allows the physician to take a picture of the whole body and locate inflammation. The investigators have found that some patients with psoriasis (but without arthritis) have inflammation in joints and tendons even before the patient has symptoms. In this study, the investigators will explore how well PET/CT works for assessing inflammation in patients with PsA. This would be a very exciting tool that could be used to find and treat inflammation before it causes damage or pain.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80,
* active psoriatic arthritis (joint or enthesis inflammation)

Exclusion Criteria:

* Diabetes,
* pregnant,
* no active PsA

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with psoriatic arthritis defined by CASPAR criteria and active joint disease.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2018-10-02 (Actual)

PRIMARY OUTCOMES:
Primary outcome is inflammation as measured by SUVmax and metabolic volumetric product in the joints and entheses. | At the discretion of the PI

SECONDARY OUTCOMES:
Correlation of local inflammation in joints and enthesis with systemic inflammatory markers including IL6 and high sensitivity CRP. | At the discretion of the PI

CONTACTS AND LOCATIONS:
Overall Officials: Alexis R Ogdie, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Division of Rheumatology, Philadelphia, Pennsylvania, United States